CLINICAL TRIAL: NCT03653364
Title: A Multicenter, Single-Arm, Open-Label Study to Assess the Safety, Pharmacokinetics, and Efficacy of Baloxavir Marboxil in Otherwise Healthy Pediatric Patients From Birth to < 1 Year With Influenza-Like Symptoms
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Efficacy of Baloxavir Marboxil in Healthy Pediatric Participants From Birth to < 1 Year With Influenza-Like Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP40559; 2018-002154-70 (EudraCT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baloxavir Marboxil (Experimental): Participants will receive single oral dose of baloxavir marboxil on Day 1 (based on body weight and age).
  Interventions: Drug: Baloxavir Marboxil

INTERVENTIONS:
Drug: Baloxavir Marboxil — Participants will receive single oral dose of baloxavir marboxil on Day 1 based on body weight and age. Participants aged ≥ 3 months to <12 months old received baloxavir marboxil, 2 milligrams per kilograms (mg/kg). Participants from birth to < 4 weeks old and ≥ 4 weeks to < 3 months old received baloxavir marboxil, 1 mg/kg.

SUMMARY:
This study will evaluate the safety, pharmacokinetics and efficacy of baloxavir marboxil in healthy pediatric participants from birth to <1 year with influenza like symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age from birth to < 1 year at screening
* Written informed consent for study participation obtained from participant's parents or legal guardian
* Parent/guardian willing and able to comply with study requirements, in the investigator's judgment
* Participants with a diagnosis of influenza virus infection confirmed by the presence of all of the following:

  1. In the investigator's judgement there is a clinical suspicion of influenza
  2. At least one respiratory symptom (either cough or coryza)

  (b) Positive prescreening influenza test (RIDT or PCR) performed within 48 hours of screening
* Participants with a negative prescreening COVID-19 test (RAT or PCR) within 48 hours of screening
* The time interval between the onset of symptoms and screening is ≤ 96 hours (the onset of symptoms is defined as the time when body temperature first exceeded 37.5°C if known, or the time when the first symptom was noticed by the parent or caregiver)

Exclusion Criteria:

* Hospitalized for complications of influenza or significant comorbidities
* Concurrent infections requiring systemic antiviral therapy at screening
* Require, in the opinion of the investigator, any of the prohibited medication during the study
* Preterm neonates (born at < 37 weeks gestation) and/or weighing < 2.5 kg at screening
* Previous treatment with peramivir, laninamivir, oseltamivir, zanamivir, or amantadine within 2 weeks prior to screening
* Immunization with a live/attenuated influenza vaccine during the 2 weeks prior to screening
* Concomitant treatment with steroids or other immuno-suppressant therapy
* Known HIV infection or other immunosuppressive disorder
* Uncontrolled renal, vascular, neurologic or metabolic disease (e.g., diabetes, thyroid disorders, adrenal disease), hepatitis, cirrhosis, or pulmonary disease or participants with known chronic renal failure
* Active cancer at any site
* History of organ transplant
* Known hypersensitivity to study drug (i.e., baloxavir marboxil) or to acetaminophen
* Participation in a clinical trial within 4 weeks or five half-lives of exposure to an investigational drug prior to screening, whichever is longer

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (8):
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Usf Health, Tampa, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago;Division of Infectious Disease, Chicago, Illinois
  - Kentucky Pediatric Research Center, Bardstown, Kentucky
  - Oak Cliff Research Company, LLC, Dallas, Texas
  - Mercury Clinical Research, Houston, Texas
  - Tekton Research, San Antonio, Texas
- Bulgaria (2):
  - MHAT Stamen Iliev AD, Montana
  - SHAT for Pneumo-Phtysiatric Diseases ?Dr. Dimitar Gramatikov?; Dept. of Pulmonology and Phtisiatrics, Rousse
- ICIMED Instituto de Investigación en Ciencias Médicas, San José, Costa Rica
- TAYS Lastenklinikka; Lasten lääketutkimuskeskus Peetu, Tampere, Finland
- Clalit Health Services- Pediatric Ambulatory Clinic; Pediatric Ambulatory Clinic, Petah Tikva, Israel
- Poland (5):
  - NZOZ Salmed, ??czna
  - Samodzielny Zespol Publicznych Zakladow Opieki Zdrowotnej im. Dzieci Warszawy w Dziekanowie Lesnym, ?omianki
  - Wojewodzki Szpital Obserwacyjno-Zakazny; Oddzia? Pediatrii, Chorób Infekcyjnych i Hepatologii, Bydgoszcz
  - IN VIVO Sp. z o.o., Bydgoszcz
  - NZOZ Vitamed, Bydgoszcz
- The scientific-research institute of epidemiology; Infectious clinical hospital ?2 of Moscow H.D., Moskva, Moscow Oblast, Russia
- South Africa (6):
  - Global Clinical Trials; Clinical Trials, Gauteng
  - GAMA; Clinical Research, Germiston
  - Peermed Clinical Trial Centre, Kempton Park
  - Metropolitan Clinical Research Institute, Polokwane
  - Pholosho Netcare; Netcare Hospital, Polokwane
  - Setshaba Research Centre; Clinical Research, Pretoria
- Spain (2):
  - Complejo Hospitalario Universitario de Santiago (CHUS); Area Asistencial Integrada de Pediatría, Santiago de Compostela, LA Coruña
  - Hospital Universitario 12 de Octubre; Servicio de Pediatria, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study at 15 investigative sites in 7 countries (Costa Rica, Finland, Mexico, Poland, South Africa, Spain, and the United States) from 23 January 2019 to 03 April 2023.
Pre-assignment Details: A total of 49 pediatric participants from birth to <1 year with influenza-like symptoms were enrolled in this study to receive baloxavir marboxil. Out of the 49 participants, one participant was screened and enrolled by accident but was not dosed.
Groups:
- Baloxavir Marboxil: Participants received a single oral dose of baloxavir marboxil on Day 1 based on body weight and age.
Period: Overall Study
Arm/Group | Baloxavir Marboxil
Started | 49
Completed | 46
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Enrolled in Error | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety-evaluable population included all participants who received at least one dose of treatment regardless of whether they had any follow-up assessments.
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: days] | 206.5 (106.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From Day 1 up to Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 48
Participants
  AEs | 23
  SAEs | 2

2. Secondary Outcome: Plasma Concentrations of Baloxavir Marboxil and S-033447
Description: S-033447 is an active metabolite of baloxavir marboxil.
Time Frame: 0.5 to 2 hours post dose on Day 1; 24 hours (Day 2) and 72 hours (Day 4) post dose, Day 6 and Day 10
Population: Pharmacokinetics (PK)-evaluable population included all participants in the ITT population who had at least one post-dose drug concentration measurement at a scheduled visit timepoint. Overall number analyzed is the number of participants with data available for analysis. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 46
nanograms per milliliters (ng/mL)
  Baloxavir Marboxil: 0.5 to 2 hours: number analyzed (Participants) | 39
  Baloxavir Marboxil: 0.5 to 2 hours | 0.93 (2.301)
  Baloxavir Marboxil: 24 hours: number analyzed (Participants) | 18
  Baloxavir Marboxil: 24 hours | 0 (0)
  Baloxavir Marboxil: 72 hours: number analyzed (Participants) | 22
  Baloxavir Marboxil: 72 hours | 0 (0)
  Baloxavir Marboxil: Day 6: number analyzed (Participants) | 27
  Baloxavir Marboxil: Day 6 | 0 (0)
  Baloxavir Marboxil: Day 10: number analyzed (Participants) | 13
  Baloxavir Marboxil: Day 10 | 0 (0)
  S-033447: 0.5 to 2 hours: number analyzed (Participants) | 39
  S-033447: 0.5 to 2 hours | 81.98 (89.412)
  S-033447: 24 hours: number analyzed (Participants) | 17
  S-033447: 24 hours | 49.75 (40.987)
  S-033447: 72 hours: number analyzed (Participants) | 22
  S-033447: 72 hours | 17.88 (17.438)
  S-033447: Day 6: number analyzed (Participants) | 27
  S-033447: Day 6 | 4.72 (3.649)
  S-033447: Day 10: number analyzed (Participants) | 13
  S-033447: Day 10 | 1.35 (1.547)

3. Secondary Outcome: Area Under the Concentration to Time Curve From Time 0 to Infinity (AUC0-inf) of Baloxavir Marboxil and S-033447
Description: S-033447 is an active metabolite of baloxavir marboxil.
Time Frame: Up to Day 10
Population: PK-evaluable population included all participants in the ITT population who had at least one post-dose drug concentration measurement at a scheduled visit timepoint. Overall number analyzed is the number of participants with data available for analysis. Since baloxavir marboxil was barely measurable in plasma, baloxavir marboxil pharmacokinetic parameters were not determined.
Measure: Mean (Standard Deviation); unit: nanograms/milliters*hour (ng/mL*hr)
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 46
nanograms/milliters*hour (ng/mL*hr)
  Baloxavir Marboxil | NA (NA) — Baloxavir marboxil was below the level of detection in plasma; hence mean and standard deviation could not be derived.
  S-033447 | 5070 (3520)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Baloxavir Marboxil and S-033447
Description: S-033447 is an active metabolite of baloxavir marboxil.
Time Frame: Up to Day 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanograms/ milliters (ng/ml)
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 46
nanograms/ milliters (ng/ml)
  Baloxavir Marboxil | NA (NA) — Baloxavir marboxil was below the level of detection in plasma; hence mean and standard deviation could not be derived.
  S-033447 | 127 (81.0)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Baloxavir Marboxil and S-033447
Description: S-033447 is an active metabolite of baloxavir marboxil.
Time Frame: Up to Day 10
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 46
hours
  Baloxavir Marboxil | NA [NA to NA] — Baloxavir marboxil was below the level of detection in plasma; hence median and full range (upper limit and lower limit) could not be derived.
  S-033447 | 4.5 [2.00 to 14.5]

6. Secondary Outcome: Apparent Half-Life (T1/2) of Baloxavir Marboxil and S-033447
Description: S-033447 is an active metabolite of baloxavir marboxil.
Time Frame: Up to Day 10
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 46
hours
  Baloxavir Marboxil | NA [NA to NA] — Baloxavir marboxil was below the level of detection in plasma; hence median and full range (upper limit and lower limit) could not be derived.
  S-033447 | 23.1 [13.0 to 33.4]

7. Secondary Outcome: Time to Alleviation of Influenza Signs and Symptoms
Description: Time to alleviation of influenza signs and symptoms was defined as the length of time taken from the start of treatment to the point at which all of the following criteria were met and remained for at least 21.5 hours:
  * A score of 0 (no problem) or 1 (minor problem) for cough and nasal symptoms for items 14 and 15 of the Canadian Acute Respiratory Illness and Flu Scale [CARIFS]);
  * A "yes" response to the following question on the CARIFS: "Since the last assessment has the participant been able to return to day care/school, or resume his or her normal daily activity in the same way as performed prior to developing the flu?";
  * First return to afebrile state (tympanic temperature ≤37.2 degree Celsius [°C]).
  Median time was estimated from the Kaplan-Meier curve. Participants who withdrew prior to an event of interest or did not experience resolution of symptoms were censored at the last observation time point.
Time Frame: Day 1 up to Day 15
Population: Intent-to-Treat Influenza-Infected (ITTi) population is a subset of ITT participants who had a laboratory confirmation of influenza infection (polymerase chain reaction [PCR] result) from any swab sample collected at baseline or during the study.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 15
hours | 163.7 [122.5 to NA] — Due to low number of participants with event, the upper limit of 95% confidence interval (CI) could not be calculated.

8. Secondary Outcome: Duration of Fever
Description: Duration of fever was defined as the length of time taken by participants to return to afebrile state [tympanic temperature ≤ 37.2°C] and remaining so for at least 21.5 hours after onset. Participants who did not have fever at baseline or whose body temperature was not collected were excluded from the analysis. Median time was estimated from the Kaplan-Meier curve.
Time Frame: Day 1 up to Day 15
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Overall number analyzed is the number of participants available for analysis.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 13
hours | 23.1 [22.3 to 44.6]

9. Secondary Outcome: Duration of Symptoms
Description: The efficacy of baloxavir marboxil was evaluated by duration of symptoms i.e., alleviation of all symptoms as defined by a score of 0 [no problem] or 1 [minor problem] and remaining so for at least 21.5 hours, for all 18 symptoms (Poor appetite; Not sleeping well; Irritable, cranky, fussy; Feels unwell; Low energy, tired; Not playing well; Crying more than usual; Needing extra care; Clinginess; Headache; Sore throat; Muscle aches or pains; Fever; Cough; Nasal congestion, runny nose; Vomiting; Not interested in what's going on; Unable to get out of bed) specified in the CARIFS questionnaire. Median time was estimated from the Kaplan-Meier curve. Participants who withdrew prior to an event of interest or did not experience resolution of symptoms were censored at the last observation time point.
Time Frame: Day 1 up to Day 15
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 15
hours | 163.7 [71.0 to NA] — Due to low number of participants with event, the upper limit of 95% confidence interval (CI) could not be calculated.

10. Secondary Outcome: Time to Return to Normal Health and Activity
Description: Time to return to normal health and activity was defined by a 'Yes' response to the following question on the CARIFS: "Since the last assessment has the patient been able to return to day care/school or resume his or her normal daily activity in the same way as performed prior to developing the flu?" and remaining so for at least 21.5 hours.
  Median time was estimated from the Kaplan-Meier curve.Participants who withdrew prior to an event of interest or did not experience resolution of symptoms were censored at the last observation time point.
Time Frame: Day 1 up to Day 15
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Overall number analyzed is the number of participants with data available for analysis
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 14
hours | 140.7 [72.2 to NA] — Due to low number of participants with event, the upper limit of 95% confidence interval (CI) could not be calculated.

11. Secondary Outcome: Number of Participants With Influenza-Related Complications
Description: The influenza related complications include death, hospitalization, radiologically confirmed pneumonia, bronchitis, sinusitis, otitis media, encephalitis/encephalopathy, febrile seizures, myositis
Time Frame: Day 1 up to Day 29
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 15
Participants | 0

12. Secondary Outcome: Number of Participants Requiring Antibiotics
Description: The number of participants who required antibiotics for influenza related complication are reported here.
Time Frame: Day 1 up to Day 29
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 15
Participants | 0

13. Secondary Outcome: Time to Cessation of Viral Shedding by Virus Titer
Description: Time to cessation of viral shedding by virus titer was defined as the time, in hours, between the initiation of any study treatment and first time when the influenza virus titer was below the limit of detection (0.75 log10 tissue culture infectious dose (TCID)50/milliliters [mL]). Participants whose virus titers did not reach the limit by the last observation time point were treated as censored at that time point. One day was converted into 24 hours. Median time was estimated from the Kaplan-Meier curve.
Time Frame: Day 1 up to Day 29
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 10
hours | 24.5 [24.2 to 68.6]

14. Secondary Outcome: Time to Cessation of Viral Shedding by Reverse Transcription-Polymerase Chain Reaction (RT-PCR)
Description: Time to cessation of viral shedding by RT-PCR, in hours, was defined as the time between the initiation of study treatment and first time when the virus ribonucleic acid (RNA) by RT-PCR qualitative result was negative (no cycle threshold [Ct]-value detectable). Participants who did not have a negative result by the last observation time point were treated as censored at that time point. For the participants with multiple virus types, this endpoint was defined as the time between the initiation of the study treatment and first time when the virus RNA by RT-PCR qualitative result was negative for all virus types. One day was converted into 24 hours. Median time was estimated from the Kaplan -Meier curve. Participants with a positive virus RNA on Day 1 are included in this analysis.
Time Frame: Day 1 up to Day 29
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Overall number analyzed is the number of participants with a positive virus RNA on Day 1.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 14
hours | 219.1 [141.6 to 695.5]

15. Secondary Outcome: Change From Baseline in Influenza Virus Titer Over Time
Description: Change from baseline in influenza virus titer (log10TCID50/mL) was defined as the change from baseline in influenza virus titer on Days 2, 4, 6, 10, and 29. If influenza virus titer was less than the lower limit of quantification (LLOQ), the virus titer was imputed as 0.749 (log10TCID50/mL). Only participants with a positive virus titer on Day 1 were included in this analysis.
Time Frame: Baseline, Days 2, 4, 6, 10, and 29
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Mean (Standard Deviation); unit: log10 TCID 50/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 15
log10 TCID 50/mL
  Baseline: number analyzed (Participants) | 10
  Baseline | 3.58 (1.81)
  Change From Baseline at Day 2: number analyzed (Participants) | 10
  Change From Baseline at Day 2 | -2.50 (1.70)
  Change From Baseline at Day 4: number analyzed (Participants) | 10
  Change From Baseline at Day 4 | -2.60 (1.95)
  Change From Baseline at Day 6: number analyzed (Participants) | 10
  Change From Baseline at Day 6 | -2.43 (1.40)
  Change From Baseline at Day 10: number analyzed (Participants) | 10
  Change From Baseline at Day 10 | -2.83 (1.81)
  Change From Baseline at Day 29: number analyzed (Participants) | 4
  Change From Baseline at Day 29 | -1.69 (1.71)

16. Secondary Outcome: Change From Baseline in the Amount of Virus RNA (RT-PCR) Over Time
Description: Change from baseline in the amount of virus RNA was defined as the change from baseline in the amount of virus RNA on Days 2, 4, 6 and 10. If the amount of virus RNA is less than the lower limit of quantification, the amount of virus RNA was imputed as the relevant LLOQ (log10 viral particles per mililiter (vp/mL)). If a participant was infected with multiple virus types, the sum of virus RNA (log10 vp/mL) was used for analysis. Participants with a positive virus RNA by RT-PCR on Day 1 were included in this analysis.
Time Frame: Baseline, Days 2, 4, 6, and 10
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log10 vp/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 15
log10 vp/mL
  Baseline: number analyzed (Participants) | 14
  Baseline | 6.46 (1.91)
  Change From Baseline at Day 2: number analyzed (Participants) | 12
  Change From Baseline at Day 2 | -2.26 (1.00)
  Change From Baseline at Day 4: number analyzed (Participants) | 12
  Change From Baseline at Day 4 | -1.93 (1.99)
  Change From Baseline at Day 6: number analyzed (Participants) | 9
  Change From Baseline at Day 6 | -1.76 (2.40)
  Change From Baseline at Day 10: number analyzed (Participants) | 6
  Change From Baseline at Day 10 | -3.30 (3.46)

17. Secondary Outcome: Percentage of Participants With Positive Influenza Virus Titer Over Time
Description: Percentage of participants positive for influenza virus titer at each visit were defined as the percentage of participants whose influenza virus titer was not less than the LLOQ (0.75 log10TCID50/mL) or positive among those assessed for influenza virus titer on Days 2, 4, 6, 10 and 29. Participants with a positive influenza virus titer on Day 1 were included in this analysis.
Time Frame: Baseline, Days 2, 4, 6, 10, and 29
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Overall number analyzed is the number of participants with a positive influenza virus titer on Day 1. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 10
percentage of participants
  Baseline | 100
  Day 2 | 40
  Day 4 | 20
  Day 6 | 30
  Day 10 | 0
  Day 29: number analyzed (Participants) | 4
  Day 29 | 0

18. Secondary Outcome: Percentage of Participants Positive by RT-PCR Over Time
Description: Percentage of participants positive by RT-PCR at each visit was defined as the percentage of participants with a positive qualitative result among those assessed by RT-PCR on Days 2, 4, 6, 10 and 29. Participants with a positive RT-PCR result on Day 1 were included in this analysis. Percentages are rounded off.
Time Frame: Baseline, Days 2, 4, 6, 10, and 29
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Overall number analyzed is the number of participants with a positive RT-PCR result on Day 1. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 14
percentage of participants
  Baseline | 100
  Day 2: number analyzed (Participants) | 13
  Day 2 | 92.3
  Day 4: number analyzed (Participants) | 13
  Day 4 | 92.3
  Day 6 | 64.3
  Day 10 | 42.9
  Day 29: number analyzed (Participants) | 7
  Day 29 | 0

19. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) in Virus Titer
Description: AUC in virus titer was calculated using the trapezoidal method. Twenty-four hours of time was converted into one day. Participants with a positive virus titer on Day 1 were included in this analysis. The LLOQ and lower limit of detection was defined as 0.75 log10TCID50/mL for flu A and 0.75 log10TCID50/mL for flu B. If a participant was infected with multiple virus types, the sum of those virus titers will be used for analysis.
Time Frame: Day 1 up to Day 29
Population: ITTi population is a subset of ITT participants who had a laboratory confirmation of influenza infection (PCR result) from any swab sample collected at baseline or during the study. Overall number analyzed is the number of participants with a positive virus titer on Day 1.
Measure: Mean (Standard Deviation); unit: log10 TCID 50/mL*hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 10
log10 TCID 50/mL*hours | 405.23 (184.72)

20. Secondary Outcome: Area Under the Curve in the Amount of Virus RNA (RT-PCR)
Description: AUC in virus RNA (RT-PCR) was defined as AUC of change from baseline in the amount of virus RNA (RT-PCR). AUC was calculated using the trapezoidal method similar to AUC in virus titer. Participants with a positive RT-PCR result on Day 1 were subjected to this analysis. If the amount of virus RNA is less than the lower limit of quantification, the amount of virus RNA was imputed as the relevant LLOQ (log10 viral particles per mililiter (vp/mL)). If a participant was infected with multiple virus types, the sum of those the amount of virus RNA was used for analysis.
Time Frame: Day 1 up to Day 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: log10 vp/mL*hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 13
log10 vp/mL*hours | 779.06 (426.83)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 29
Description: Safety-evaluable Population included all participants who received at least one dose of treatment regardless of whether they had any follow-up assessments.
Arm/Group | Baloxavir Marboxil
All-Cause Mortality (participants affected / at risk) | 1/48
Serious Adverse Events (participants affected / at risk) | 2/48
Other Adverse Events (participants affected / at risk) | 11/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baloxavir Marboxil (N=48)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baloxavir Marboxil (N=48)
Diarrhoea (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 6 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT03653364/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03653364/SAP_001.pdf